CLINICAL TRIAL: NCT07179549
Title: Evaluation of the Incidence of Myocardial Damage Following Upper and Lower Gastrointestinal Endoscopy in High-risk Patients: MINS-Endoscopy Study
Brief Title: Evaluation of the Incidence of Myocardial Damage Following Upper and Lower Gastrointestinal Endoscopy in High-risk Patients
Status: Not yet recruiting | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: MINS-Endoscopy Study
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: GI Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypoperfusion occurs following anaesthesia induction as a result of:

1. a reduction in venous return and cardiac output subsequent to the dilatation of the venous reservoir, and
2. a reduction in mean arterial pressure (MAP) secondary to arteriolar vasodilatation (reduction in arterial resistance) and decreased cardiac output. Many studies in the literature have focused on intraoperative hypotension and have reported an association between intensity x duration of hypotension and the occurrence of postoperative adverse events. Smaller interventional studies have suggested that improving stroke volume (SV, and therefore cardiac output) using fluid titration could reduce postoperative complications. Among postoperative adverse events consecutive to hypoperfusion, the occurrence of myocardial injury after noncardiac surgery (MINS) is well documented and is correlated to postoperative mortality at day 30.

Upper and lower gastro-intestinal (GI) endoscopies are frequently performed under sedation (i.e.: general anaesthesia without orotracheal intubation) as daycare procedures. More than 10% of all anaesthesia worldwide is administered for GI endoscopic procedures. A substantial proportion of patients undergoing these procedures have significant comorbidities, classifying them as ASA 3 or ASA 4. However, despite the higher risk associated to their comorbidities, these patients are most often monitored intraoperatively as if they were ASA 1 or ASA 2, i.e.: using intermittent oscillometric blood pressure measurements every 5 minutes, an electrocardioscope and peripheral oxygen saturation measurement. They are also usually considered eligible for daycare procedures. However, hypoperfusion occurs during upper and lower GI endoscopies as a result of anaesthesia combined with abdominal insufflation (stomach followed by colon) and always starts with a decrease in SV, followed by a decrease in MAP.

The exact incidence of MINS following endoscopic procedures in high-risk patients has not been investigated to our knowledge and is not known precisely. The first part of this pragmatic study would consist in collecting pre-op and post-op (4 hours post procedure) plasma troponin level in ASA 3 or ASA 4 patients scheduled for upper and lower GI endoscopy at the time of routine blood collection. The patient will also be monitored using a Clearsight® continuous hemodynamic monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients scheduled for upper and lower GI endoscopy
* ASA class 3 or 4: patients considered by anesthesiologists at "high risk" of postoperative complications, based on their comorbidities

Exclusion Criteria:

* Symptomatic coronary artery disease at the time of inclusion
* Pulmonary embolism less than two weeks before inclusion
* Septic shock less than two weeks before inclusion
* Patients with renal failure, with glomerular filtration rate<40 ml/min
* Patient not covered by social security
* Patient is pregnant
* Protected Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients considered high risk
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ultra-sensitive Troponin I plasma level | 4 hours
  Ultra-sensitive Troponin I plasma level variation following upper and lower GI endoscopy. Troponin I will be measured immediately prior to anaesthesia induction (IV line placement) and before patient discharge of the hospital, i.e.: 4 (±1) hours after the procedure.
Ultra-sensitive Troponin I plasma level variation following upper and lower GI endoscopy. | 4 hours
  Ultra-sensitive Troponin I plasma level variation following upper and lower GI endoscopy. Troponin I will be measured immediately prior to anaesthesia induction (IV line placement) and before patient discharge from the hospital, i.e.: 4 (±1) hours after the procedure

IPD SHARING:
Plan to Share IPD: No
privacy, ethical, or regulatory reasons